CLINICAL TRIAL: NCT00432484
Title: Lingzhi (Ganoderma Lucidum) and Sen Miao San Supplementation in Rheumatoid Arthritis(RA): An Animal Model and A Phase I Study
Brief Title: Lingzhi and Sen Miao San for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Lai-Shan Tam, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-2005-001
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Lingzhi; Sen Miao San; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Placebo Comparator): Placebo with Lingzhi(Granoderma Lucidum) and Sen Miao San
  Interventions: Drug: Lingzhi and Sen Miao San

INTERVENTIONS:
Drug: Lingzhi and Sen Miao San — G lucidum and SMS were supplied as capsules, containing 4.0 gm of G lucidum extract, 2.4 gm of Rhizoma atractylodis (Cangzhu), 2.4 gm of Cotex phellodendri(Huangbai), and 2.4 gm of Radix achyranthes Bidentatae(Niuxi). Each patient took either 3 capsules twice daily as recommended by the TCM experts or identical-looking placebo.
  Other Names: Pingyin English name; Lingzhi Ganoderma lucidum seu Japonicum; Cangzhu Atractylodes lancea; Huangbo Phellodendron amurense; Niuxi Achyranthes bidentata B1

SUMMARY:
To study the efficacy of TCM as an effective supplement in addition to the traditional treatment in RA.

DETAILED DESCRIPTION:
It is a prospective, double-blind, randomized, placebo-controlled study in patients with RA. It consists of a 24 - weeks period of randomized double-blind treatment of either TCM(Lingzhi and Sen Miao San)or placebo.

Primary outcome is assessed by showing a clinical response of at least 20% and 50% as defined by the American College of Rheumatology (ACR) criteria.Secondary outcome is defined as the changes in the number of swollen and tender joint counts, and the levels of ESR, CRP, the inflammatory markers, cytokine levels and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the 1987 American College of Rheumatology (ACR) criteria for RA.
* The presence of 2 or more swollen or tender joints, based on 28-joint count.
* Morning stiffness lasting for 30 minutes.
* Erythrocyte sedimentation rate (ESR) of 28 mm/hour, despite treatment with disease modifying agent including MTX, sulphasalazine, hydroxychloroquine, auranofin or azathioprine were recruited into the study.
* Patients taking glucocorticoids (prednisone < 7.5 mg/day) and/or nonsteroidal antiinflammatory drugs must have been taking a stable dosage for at least 4 weeks before entering the trial and were required to take the same dosage throughout the trial.
* Patients had radiographic erosive diseases.

Exclusion Criteria:

* Patients who are pregnant or nursing mothers.
* Severe liver disease (e.g cirrhosis, chronic active hepatitis)
* Renal impairment (serum creatinine level > 150mmol/L)
* Known hypersensitivity to herbal medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
We assessed the proportion of patients showing a clinical response of at least 20% and 50% as defined by the American College of Rheumatology (ACR) criteria (20). | wk52

SECONDARY OUTCOMES:
The change in the number of swollen and tender joint counts, and the levels of ESR, CRP, the inflammatory markers, cytokine levels and oxidative stress will be assessed as secondary outcomes. | wk52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Institute of Chinese Medicine, Hong Kong, China

REFERENCES:
- [Derived] Li EK, Tam LS, Wong CK, Li WC, Lam CW, Wachtel-Galor S, Benzie IF, Bao YX, Leung PC, Tomlinson B. Safety and efficacy of Ganoderma lucidum (lingzhi) and San Miao San supplementation in patients with rheumatoid arthritis: a double-blind, randomized, placebo-controlled pilot trial. Arthritis Rheum. 2007 Oct 15;57(7):1143-50. doi: 10.1002/art.22994. PMID 17907228